CLINICAL TRIAL: NCT06151483
Title: Intensive Versus Standard Treatment for Spinal Anesthesia-induced Hypotension on Maternal and Neonatal Outcomes During Cesarean Section: A Multicenter, Prospective, Single-blind, Randomized, Controlled Trial
Brief Title: Intensive Versus Standard Treatment for Spinal Anesthesia-induced Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Yi Chen-2024-1
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2023-12

CONDITIONS: Outcome
MeSH Terms: interventions — Vasoconstrictor Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (Active Comparator): The maternal systolic blood pressure was consistently maintained above 80% of the preoperative baseline value from the initiation of spinal anesthesia until fetal delivery.
  Interventions: Drug: Alpha-Agonist
- Intensive group (Experimental): The maternal systolic blood pressure was consistently maintained above 90% of the preoperative baseline value from the initiation of spinal anesthesia until fetal delivery.
  Interventions: Other: α-adrenergic receptor agonist

INTERVENTIONS:
Drug: Alpha-Agonist — The maternal systolic blood pressure was consistently maintained above 80% of the preoperative baseline value from the initiation of spinal anesthesia until fetal delivery.
  Other Names: Vasopressors
  Arms: Standard group
Other: α-adrenergic receptor agonist — The maternal systolic blood pressure was consistently maintained above 90% of the preoperative baseline value from the initiation of spinal anesthesia until fetal delivery.
  Other Names: Vasopressors
  Arms: Intensive group

SUMMARY:
The objective of this study is to investigate the impact of varying maternal blood pressure maintenance targets on neonatal outcomes following cesarean section.

DETAILED DESCRIPTION:
Post-spinal anesthesia hypotension is a frequent complication during spinal anesthesia for cesarean section. The incidence of post-spinal anesthesia hypotension is as high as 62.1-89.7% if prophylactic measures are not taken. The 2016 ASA guidelines for obstetric anesthesia suggest avoiding hypotension following spinal anesthesia in women and emphasize the use of vasopressors, specifically alpha-receptor agonists, as the preferred strategy to prevent and manage post-spinal anesthesia hypotension. The 2018 International Consensus in the United Kingdom and Northern Ireland recommends maintaining maternal systolic blood pressure above 90% of the baseline value following lumbar anesthesia, while avoiding dropping below 80% of the baseline value. Currently, the threshold for maintaining blood pressure above 80% of the baseline value is widely adopted as a standard; however, limited evidence supports the advantage of sustaining maternal blood pressure above 90% of the baseline value. The objective of this study is to investigate the impact of varying maternal blood pressure maintenance targets on neonatal outcomes following cesarean section.

ELIGIBILITY:
Criteria: Inclusion Criteria:

* 18-45 years
* Primipara or multipara
* Singleton pregnancy ≥37 weeks
* American Society of Anesthesiologists physical status classification I to II
* Scheduled for cesarean section under spinal anesthesia

Exclusion Criteria:

* Body height < 150 cm
* Body weight > 100 kg or body mass index (BMI) ≥ 40 kg/m2
* Eclampsia or chronic hypertension or baseline blood pressure ≥180 mmHg
* Hemoglobin < 7g/dl
* Fetal distress, or known fetal developmental anomaly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1184 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
pH | Immediately after delivery
  From umbilical arterial blood gases.
Base excess | Immediately after delivery
  From umbilical arterial blood gases.

SECONDARY OUTCOMES:
The incidence of post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 80% of the baseline
The incidence of severe post-spinal anesthesia hypotension. | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 60% of the baseline.
The incidence of bradycardia. | 1-15 minutes after spinal anesthesia
  Heart rate < 50 beats/min.
The incidence of nausea and vomiting. | 1-15 minutes after spinal anesthesia
  Presence of nausea and vomiting in patients after spinal anesthesia
The incidence of hypertension. | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) >120% of the baseline.
Partial pressure of oxygen (PO2) | Immediately after delivery
  From umbilical arterial blood gases.
APGAR score | 1 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration; 0(Worst)-10(Best)
APGAR score | 5 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration; 0(Worst)-10(Best)

CONTACTS AND LOCATIONS:
Overall Officials: Xinli Ni, M.D., Study Chair — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China